CLINICAL TRIAL: NCT02602756
Title: Phase II Trial, Randomized, Under Single-blind Conditions, Assessing Two Models of Modified Hypofractionated Proton-therapy on Patients With Large Choroidal Melanomas
Brief Title: Study Assessing Two Models of Hypofractionated Protontherapy on Large Choroidal Melanomas
Acronym: HYGROMEL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient quality of data collection
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/02
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Melanoma
Keywords: Choroid Melanoma
MeSH Terms: conditions — Melanoma; Uveal Melanoma

STUDY DESIGN:
Intervention Model Description: Study with 2 differents dosages of proton therapy
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Protontherapy : 4 sessions of 13 Gy, total dosis 52 Gy
  Interventions: Radiation: Protontherapy
- B (Experimental): Protontherapy : 8 sessions of 6.5 Gy, total dosis 52 Gy
  Interventions: Radiation: Protontherapy

INTERVENTIONS:
Radiation: Protontherapy — Proton-therapy consists in four consecutive sessions. The experimental arm consists in eight sessions. Irradiation is administered over two weeks, delivering a total dose of 60 Cobalt Gris Equivalent (CGE is the physical Gray dose multiplied by a biological factor of relative efficiency of 1.1 for protons compared to photons).

SUMMARY:
Ocular melanomas have been treated for a long time by enucleation, with an unfavorable major impact on the patient's quality of life, social life, self-image, how they feel about others and about living with this disability. As a matter of fact, classical radiation therapy by photons is not accurate enough to deliver a sufficiently high dose to eradicate a melanoma without causing irreversible ocular brain complications since these tumors are " relatively radio resistant ". The possibility of delivering high doses due to the precision of protons ("Bragg peak") has allowed to overcome this limitation. The conservative uveal melanoma treatment has become a standard after the Collaborative Ocular Melanoma Study (COMS) indicating an equivalent rate of metastases and a non-impaired survival rate with a conservative treatment when compared to immediate enucleation. The quality of life benefits due to a conservative treatment has been demonstrated. Protontherapy dose has been defined in an empirical manner, it is probably excessive even if it applies to radio-resistant tumors. In France, radiotherapy by protons for choroidal melanomas delivers a dose of 60 Gy cobalt equivalent (that is 52 measured Gy, or " Physical dose") in 4 fractions and 4 days.

Referential treatment of ocular melanomas (other than conjunctiva) indicates proton-therapy for T1, T2, T3 < 40% of ocular volume, and T4 only if extra scleral extension ≤ 2mm. However, there is an enucleation indication for T3 > 40% of ocular volume and T4.

Our purpose is to override this relative contraindication, choroidal melanoma volume ≥ 40% of ocular volume. As a matter of fact, the investigators observe an increasing demand from ophthalmologists and patients for not performing primary enucleation. Also, during the last five years treatment of complications have improved and a less " hard " hypo fractionation (6.5 Gy per fraction) has equivalent local control results as for " hard " fractionation (13 Gy per fraction).

DETAILED DESCRIPTION:
A more fractioned proton-therapy treatment, with doses per fraction of 6.5 Gy rather than 13 Gy, can limit the rate and the severity of complications degrading the quality of life by complications (pain, diminished visual acuity) and treatments (intra-ocular injections...).

In this study, patients will receive a total dose of 52 Gy in four 13 Gy sessions for the standard arm and in eight 6.5 Gy sessions for the experimental arm.

The investigators expect an identical local control rate within 2 year's time with a decrease in rate and severity of severe complications due to adapted fractionation (eight sessions with lower doses instead of four fractions with very high doses as it is usually recommended in the guidelines for small to medium melanomas).

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with choroidal melanoma by an ophthalmologist and proton-therapy treatment proposed by the multi-disciplinary board meeting
* Patient over 18 years old, male or female
* Performance status ≤ 2
* Size and/or thickness greater than those proposed on proton-therapy appendix indications (tumor volume/ocular globe > 40% and/or thickness ≥ 12 mm and/or diameter ≥ 18 mm or thickness ≥ 10 mm and diameter ≥ 15 mm). Possible ophthalmological follow-up examinations at 6 months, one year, 18 months and two years.
* No contraindication for adjuvant chemotherapy
* Authorized technique to preserve the optic nerve
* Patient having undergone the required medical procedures:

  * Ophthalmological examination
  * Clip positioning
  * Proton-therapy treatment (localization CT, first simulation, second simulation, final simulation)
* Patient reads information note and signs consent form

Exclusion Criteria:

* Exclusive iris damage
* Exclusive conjunctival damage
* First melanoma surgery
* Enucleation planned post-proton-therapy
* Exentration indication
* Life expectancy < 2 years
* Scleral exteriorisation > 2 mm
* Absolute radiotherapy contraindication (ataxia-telangiectasia)
* Cancer history, except for complete remission cancers of over 5 years, basocellular skin carcinomas completely resected, in-situ carcinomas or treated in situ cervical epithelioma
* Presence of metastases other than hepatic (endoresection authorized)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
local control rate without severe complications 2 years after. | up to 60 months

SECONDARY OUTCOMES:
Enucleation rate | up to 60 months
Tumoral transretinien endoresection by unplanned vitrectomy in inclusion (emergency procedure) | up to 60 months
Number of months without metastases evaluation | up to 60 months
Number of months of Specific global survival evaluation | up to 60 months
Complications and toxicity evaluation (number of subjects with adverse events related to treatment) | up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Juliette THARIAT, md, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France

REFERENCES:
- See also: Related Info — http://www.centreantoinelacassagne.org